CLINICAL TRIAL: NCT00186290
Title: Fractionated Total Body Irradiation (FTBI), Etoposide (VP-16) and Cyclophosphamide (CY) Followed by Allogeneic Bone Marrow Transplantation for Patients With Advanced Leukemia or High Grade Lymphoma
Brief Title: Allo BMT in Advanced Leukemia or High Grade Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Robert Lowsky, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT34; 74165; BMT34; NCT00186290
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia; Blood and Marrow Transplant (BMT); Lymphomas: Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia

INTERVENTIONS:
Procedure: ablative allogeneic hematopoietic cell transplantation

SUMMARY:
To evaluate the role of ablative allogeneic hematopoietic cell transplantation in the treatment of advanced leukemia or lymphoma.

DETAILED DESCRIPTION:
To determine the disease free survival and overall survival of patients with ALL and ANLL after induction failure, in relapse, or subsequent remission from CML in several phases or recurrent lymphoblastic lymphoma who receive fractionated TBI, etoposide and cyclophosphamide followed by allogenic bone marrow grafting from histocompatible sibling donors. Fractionated Total Body Irradiation (FTBI), Etoposide (VP-16) and Cyclophosphamide (CY) Followed by Allogeneic Bone Marrow Transplantation for Patients with Advanced Leukemia or High Grade Lymphoma

ELIGIBILITY:
Inclusion Criteria:HLA identical donor

* adequate organ function
* other life threatening disease

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Estimated)
Dates: Start 1989-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
overall survival | october 2009
disease free survival | October 2009

SECONDARY OUTCOMES:
early and late toxicities of the treatment regimen | October 2009

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States